CLINICAL TRIAL: NCT00731250
Title: A Randomised, Double-blind, Placebo-controlled Study to Assess the Effect of Oral, Single Dose SB-705498 in a Validated Intranasal Capsaicin Challenge Model in Healthy Volunteers
Brief Title: A Study To Assess The Effect Of SB-705498 In A Capsaicin Challenge Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 111611
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Rhinitis
Keywords: Capsaicin challenge
MeSH Terms: conditions — Rhinitis | interventions — SB 705498

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- PART 1-Visit 1-Placebo (Placebo Comparator): Eligible subjects will receive matching placebo tablets
  Interventions: Drug: Placebo
- PART 1-Visit 1-Capsaicin (Experimental): Eligible subjects will receive incremental capsaicin doses
  Interventions: Other: Caspaicin
- PART 1-Visit 2-Placebo (Placebo Comparator): Eligible subjects will receive matching placebo tablets
  Interventions: Drug: Placebo
- PART 1-Visit 2-Capsaicin (Experimental): Eligible subjects will receive maximum capsaicin dose
  Interventions: Other: Caspaicin
- PART 1-Visit 3-Placebo (Placebo Comparator): Eligible subjects will receive matching placebo tablets
  Interventions: Drug: Placebo
- PART 1-Visit 3-Capsaicin (Experimental): Eligible subjects will receive matching placebo tablets incremental capsaicin doses
  Interventions: Other: Caspaicin
- PART 2-Visit 1-Placebo (Placebo Comparator): Eligible subjects will receive matching placebo tablets
  Interventions: Drug: Placebo
- PART 2-Visit 1-SB-705498 (Experimental): Eligible subjects will receive SB-705498 tablets
  Interventions: Drug: SB-705498
- PART 2-Visit 2-Capsaicin (Experimental): Eligible subjects will receive matching placebo tablets incremental capsaicin doses
  Interventions: Other: Caspaicin

INTERVENTIONS:
Drug: SB-705498 — Subjects will be administered a single dose of 400 mg SB-705498
  Arms: PART 2-Visit 1-SB-705498
Drug: Placebo — Subjects will be administered SB-705498 matching placebo tablets
  Arms: PART 1-Visit 1-Placebo; PART 1-Visit 2-Placebo; PART 1-Visit 3-Placebo; PART 2-Visit 1-Placebo
Other: Caspaicin — Subjects will be challenged with 0.5 µg, 5.0 µg and 50 µg intranasal dose
  Arms: PART 1-Visit 1-Capsaicin; PART 1-Visit 2-Capsaicin; PART 1-Visit 3-Capsaicin; PART 2-Visit 2-Capsaicin

SUMMARY:
This study is designed to look at the affect of SB-705498 on rhinitis symptoms, as induced by capsaicin challenge

ELIGIBILITY:
Inclusion Criteria:

* Healthy.
* Male or female between 18 and 60 years of age inclusive.
* Non-child bearing women or women of child bearing potential if they agree to use contraception as indicated by the protocol
* Non-smoker for at least 6 months with a pack history <5 pack years (Pack years = (No. of cigarettes smoked/day/20) x No. of years smoked).
* Body weight > 50 kg and body mass index (BMI) within the range 19 - 29.9 kg/m2 (inclusive).
* Capable of giving written informed consent.
* Available to complete all the required study measurements.
* Normal 12-lead ECG at screening.
* For Part 2 only: The subject must demonstrate reactivity to unilateral, intranasal challenge with the selected single dose of capsaicin, defined as development of TSS ≥ 3.

Exclusion Criteria:

* Past medical history of rhinitis, including allergic, non-allergic rhinitis and rhinosinusitis.
* Nasal conditions likely to affect the outcome of the study, i.e. nasal septal perforation, nasal polyps, other nasal malformations.
* A history of gastrointestinal, hepatic, renal or multiple cardiovascular risk factors.
* Positive pre-study drug/alcohol screen.
* Positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for human immunodeficiency virus (HIV) antibody (if determined by the local standard operating procedures (SOPs)).
* History of regular alcohol consumption within 6 months of the study.
* Exposure to more than four new chemical entities within 12 months prior to the start of the study.
* Participation in a clinical trial with a new molecule entity or any other clinical trial within 4 months of the start of the study.
* Use of prescription or non-prescription drugs, as well as of vitamins, herbal and dietary supplements (including St John's Wort) within 2 days prior to each study visit in Part 1 of the study or 14 days prior to the first treatment administration in Part 2 of the study.
* Inability to abstain from all intranasal or oral medication to treat nasal symptoms from the first capsaicin challenge to the completion of the study including: sodium cromoglycate, antihistamines, anticholinergics, alpha-adrenergic agonists and corticosteroids
* History of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation.
* Subjects demonstrating hypersensitivity to the placebo capsaicin challenge at baseline screening.
* Donation of blood or blood products in excess of 500mL within a 56 day period prior the start of Part 2 of this study.
* Pregnant females as determined by positive serum or urine human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Nicotine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* For Part 2 only: Subjects with known lactose intolerance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2008-07-22 (Actual); Primary Completion 2009-03-01 (Actual); Study Completion 2009-03-31 (Actual)

PRIMARY OUTCOMES:
Symptom scores and secretion weights | up to 83 days

SECONDARY OUTCOMES:
Peak nasal inspiratory flow changes after challenge | up to 83 days
Biomarkers levels in the nasal samples | up to 83 days
Blood levels of drug | up to 83 days
Pharmacodynamic response | up to 83 days
Safety parameters | up to 83 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 111611 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/111611?search=study&search_terms=111611#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 111611 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111611 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111611 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111611 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111611 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111611 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111611 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register